CLINICAL TRIAL: NCT00611949
Title: EPT 101: New Geranium Oil Formulation for the Treatment of Neuropathy Pain
Brief Title: Comparison of 2 Vials of Components of a Synthetic Geranium Oil
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pennington Biomedical Research Center (Other)
Responsible Party: Principal Investigator, Frank Greenway, Clinical Medical Doctor, Pennington Biomedical Research Center
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: PBRC 21013; EPT 101
Record Dates: First submitted 2008-01-29; First posted 2008-02-11 (Estimated); Last update posted 2015-12-18 (Estimated); Status verified 2015-12

CONDITIONS: Neuropathic Pain
Keywords: Geranium oil; Neuropathy; Shingles; Herpes zoster
MeSH Terms: conditions — Neuralgia; Herpes Zoster

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 Geranium Oil (Active Comparator)
  Interventions: Other: Geranium oil
- 2 Geramium Oil (Active Comparator)
  Interventions: Other: Geranium oil

INTERVENTIONS:
Other: Geranium oil — 2 applications of topical oil per week for 2 weeks

SUMMARY:
The purpose of this study is to determine which component of an artificial geranium oil helps to reduce your neuropathy pain.

DETAILED DESCRIPTION:
EPT 101 is a double-blind successive crossover study designed to determine which components of a synthetic geranium oil provide analgesic relief, with the objective of identifying and purifying the active substance. This is not a hypothesis-generating trial, nor is it confirming a hypothesis. The trial uses human volunteers in an efficacy-directed decomposition of a complex mixture.

Patients with a diagnosis of neuralgia or neuropathy who respond to geranium oil will test two vials of components of a synthetic geranium oil for application to the maximally painful area in succession. They will treat their condition in the clinic and fill out a patient diary on separate days. The primary objective is the patient opinion of which vial has greatest analgesic efficacy. Efficacy will be measured primarily by reduction in pain intensity summed over the first two hours, compared with the pain intensity during the 30 minutes preceding application.

Following the comparison of the first two vials, the vial judged efficacious will be decomposed into two further vials and the patients will repeat the evaluation described above. At least eight pair-wise comparisons will be required to determine and confirm which of the 100+ ingredients of a synthetic geranium oil are analgesic, provided there is only one such ingredient.

ELIGIBILITY:
Inclusion Criteria:

* You are eligible to participate in this study if you have completed the study EPT 100 and geranium oil relieves your neuropathy pain successfully.

Exclusion Criteria:

* You are ineligible to participate in this study if you have completed the study EPT 100 and geranium oil does not relieve your neuropathy pain successfully

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2002-05; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Pain relief | 2 hrs. post-application

SECONDARY OUTCOMES:
Response to therapy at one hour, defined as reduction of pain summed over the first hour, compared between the two oils. | 1 hr. post-application

CONTACTS AND LOCATIONS:
Overall Officials: Frank Greenway, MD, Principal Investigator — Pennington Biomedical Research Center
Locations (1):
- Pennington Biomedical Research Center, Baton Rouge, Louisiana, United States